CLINICAL TRIAL: NCT06906614
Title: Analysis of Predictors of Stress Reactions in Medical Students During Simulation-Based Training
Brief Title: Psychophysiological Stress Response in Medical Students During Simulation-Based Communication Training -Study Protocol
Acronym: SIMU2025
Status: Not yet recruiting | Type: Observational
Sponsor: Masaryk University (Other)
Collaborators: Simulation Centre of the Faculty of Medicine of Masaryk University (Unknown); Department of Simulation Medicine, Faculty of Medicine, Masaryk University (Unknown)
Responsible Party: Principal Investigator, Miroslav Světlák, Department head (Department of Medical Psychology and Ethics), Masaryk University
Other Study IDs: SIMU2025
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Stress
Keywords: Medical Student Stress; Simulation-Based Training; Psychological Predictors of Stress; Physiological Stress Responses; Heart Rate Variability (HRV); Patient Communication Skills; Resilience and Self-Efficacy; High-Fidelity Simulation; Stress Management in Medical Education; Psychometric Assessments in Training

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 3rd-Year Medical Students in Simulation Training: This cohort consists of 3rd-year medical students enrolled in the Medical Psychology and Psychosomatics course, participating in simulation-based communication training.
  Interventions: Behavioral: Simulation-Based Communication Training

INTERVENTIONS:
Behavioral: Simulation-Based Communication Training — In our study, the intervention is more of an experimental situation - a scenario.
  High-fidelity scenarios include patients played by real actors displaying anxiety, aggression, silence, and emotional distress in various clinical situations such as delivering serious news or frustration for waiting for physicians. The average time of each simulation is 12 minutes.

SUMMARY:
In this study, researchers will examine key predictors of stress reactions in medical students participating in simulation-based communication training. By using psychometric questionnaires and physiological measurements, the study will assess how psychological traits, resilience, and self-efficacy impact stress responses during simulated patient interactions. These simulations use live actors to portray emotionally challenging scenarios, such as communicating with anxious or aggressive patients. The results aim to identify factors that contribute to heightened stress, ultimately guiding the development of targeted stress-management strategies to improve students' readiness for real-world clinical settings.

DETAILED DESCRIPTION:
Aims of the Study and Main Hypotheses

The primary aim of the study is to identify key predictors of stress responses in third-year medical students during simulation-based communication training. In this context, "stress" is operationalized both through continuous physiological measurements-principally heart rate variability (HRV) recorded via Polar chest bands-and through a battery of psychometric assessments. The study is designed to evaluate:

Primary Aim:

To determine the predictive value of psychological traits (e.g., resilience, self-efficacy) on physiological stress markers (e.g., HRV stability) and subjective stress ratings during high-fidelity patient interactions with live actors.

Hypothesis: Students exhibiting higher levels of resilience and self-efficacy will demonstrate lower physiological stress responses (i.e., more stable HRV) and report lower subjective stress.

Comparison of Stressors Across Scenarios:

To examine whether different simulated patient interactions-such as those involving anxious, aggressive, silent, or emotionally distressed patients-elicit distinct stress responses. This component will allow for the evaluation of scenario-specific stress effects, which could have implications for tailoring simulation training.

Influence of Personality Traits:

To investigate how personality characteristics, particularly neuroticism and extraversion, influence the magnitude of stress responses during simulations. This analysis will provide insight into the extent to which individual differences moderate stress levels.

Practical Application:

To inform the development of targeted interventions, such as tailored stress management or coping programs, specifically designed for students who are identified as being highly reactive to stress during simulations.

Study Design and Methodology

The study employs an observational cohort design. Data will be collected from third-year medical students enrolled in the Medical Psychology and Psychosomatics course, who participate in simulation-based patient interactions. The detailed methodological framework is as follows:

Data Collection Phases:

Phase 1 (Baseline): Two days prior to simulation sessions, participants will complete a comprehensive set of psychometric questionnaires to assess baseline levels of stress, anxiety, resilience, and self-efficacy.

Phase 2 (Pre-Simulation): Immediately before the simulation begins, students will fill out a pre-simulation questionnaire aimed at capturing their immediate stress and anxiety levels.

Phase 3 (Post-Simulation): Directly after the simulation, a post-simulation questionnaire will be administered to record acute stress responses.

Phase 4 (Post-Debriefing): Following the debriefing session, students will complete a final set of questionnaires to assess any changes in stress levels after reflective processing.

Physiological Monitoring:

Throughout the simulation, continuous HRV data will be collected using Polar chest bands. These devices provide objective, high-resolution data on the autonomic responses of students during live interactions with standardized patients.

Additionally, each simulation session will be supplemented by observational assessments provided by trained actors (standardized patients), focusing on indicators such as body language, communication style, and overall stress manifestation.

Outcome Measures While the primary outcomes relate to physiological markers (HRV) and subjective stress ratings, secondary outcomes will explore the moderating effects of personality traits and the impact of different scenario types on stress responses. These outcomes will serve as predictors for tailoring future simulation-based interventions, ensuring that the training environment can be optimized to both challenge students and support their learning effectively.

ELIGIBILITY:
Inclusion Criteria

* Enrollment as a 3rd-year medical student at the Faculty of Medicine, Masaryk University.
* Participation in the Medical Psychology and Psychosomatics course.
* Active involvement in simulation-based communication training sessions.
* Signed informed consent provided before the start of the study.
* Willingness to wear physiological monitoring devices (e.g., chest strap) during simulations.

Exclusion Criteria

* Inability or unwillingness to complete all phases of data collection, including pre- and post-simulation assessments.
* Absence of a smartphone with Bluetooth connectivity.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of 3rd-year medical students at the Faculty of Medicine, Masaryk University, enrolled in the Medical Psychology and Psychosomatics course. These students will participate in simulation-based communication training involving high-fidelity patient interactions with live actors. The focus is on assessing psychological and physiological stress responses to emotionally challenging patient scenarios, aiming to identify key predictors of stress and improve future training interventions.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in heart rate variability (HRV) using HR band Polar H10 | 2,5 hours during each simulation
  The primary outcome is the change in physiological stress markers, specifically heart rate variability (HRV), measured continuously during each simulation scenario. This measure assesses the immediate physiological response to stress-inducing patient interactions.The obtained data will be processed using time-domain HRV parameters - RMSSD, SDNN, pNN50 and Power Spectrum density HRV parameters - LF power, HF power, and LF/HF ratio.
State-Trait Anxiety Inventory X-II | 2 days before first simulation
  For measuring anxiety, the State-Trait Anxiety Inventory was used, which assesses both the temporary state of anxiety (state anxiety, STAI X-I) and the long-term trait anxiety (STAI X-II). In this study, the focus was placed on the STAI X-II section, which contains 20 items (items 21 to 40). Respondents rate their answers on a scale from 1 ("almost never") to 4 ("almost always"). During scoring, some items are reverse-scored, and the total score is obtained by summing all responses, with a higher score indicating a higher level of trait anxiety.
Affective Circumplex | 5 minutes before the simulation
  The Affective Circumplex is a questionnaire designed to subjectively assess emotions and self-confidence in the context of a simulation. Within this tool, respondents rate their level of competence - between the poles of "I feel competent" (have the knowledge and skills necessary for the simulation) and "I do not feel competent" (do not have the knowledge and skills necessary for the simulation). The questionnaire also includes an assessment of current emotional state, with participants choosing between the poles of "uncomfortable" and "pleasant" and between the poles of "calm" and "upset". Next, respondents rate their sense of control over their emotions, and are asked to express whether they are in control of their emotions or whether they are losing control. Finally, participants are asked to verbally express their current emotion - in one word or a short sentence, for example, "sadness", "shame" or "joy".
NASA Task Load Index (NASA-TLX) | 5 minutes after the simulation
  The NASA Task Load Index (NASA-TLX) is a tool to subjectively assess cognitive and emotional load during a simulation. Students rate six dimensions: mental and physical demands, time pressure, performance, effort, and frustration. Each dimension is assessed on a scale of 0-100, where a higher value indicates a higher burden. The NASA-TLX total score can be calculated as the average of all dimensions or using weighted scoring. This tool helps to compare students' subjective stress with objective physiological indicators of stress.

SECONDARY OUTCOMES:
Toronto Empathy Questionnaire | 2 days before first simulation
  This questionnaire is a shortened version of the original 16-item instrument, with the seven most relevant items (TEQ1, TEQ2, TEQ3, TEQ4, TEQ5, TEQ14 and TEQ16) selected for the study. Respondents answer on a Likert scale, where a value of 0 indicates "never" and a value of 4 indicates "always". The total score is obtained by summing all responses, with reverse scoring for negatively worded items before summing. A higher score indicates a higher level of empathy.
The Brief Resilience Scale | 2 days before first simulation
  An instrument designed to measure psychological resilience, the ability to recover quickly from difficult or stressful situations. The questionnaire contains 6 items, with respondents rating their answers on a scale from 1 ('strongly disagree') to 5 ('strongly agree'). When scoring, items 1, 3 and 5 are positively worded, while items 2, 4 and 6 are reverse scored. The final score is determined as the average of all responses, with a higher average indicating a higher level of psychological resilience.
General Self-Efficacy Scale (GSE) | 2 days before first simulation
  This questionnaire measures an individual's general self-confidence in solving problems and coping with challenges. It contains 10 items, all of which are positively worded. Respondents answer on a scale from 1 ("not at all valid") to 4 ("absolutely valid"). A total score is obtained by summing the scores of all responses, and higher final scores correspond to higher perceived self-efficacy.
Perceived Stress Scale (PSS) | 2 days before first simulation
  The Perceived Stress Scale (PSS) is a classic stress assessment instrument. The questions in this scale ask about feelings and thoughts during the last month. Each question has five response options ranging in value from null to four (0=never; 1=almost never; 2=sometimes; 3=fairly often; 4=very often). To find the total raw score, sum the values of the response to each question (reverse code items 4, 5, 7a and 8). Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
The Big Five Inventory-10 (BFI-10) | 2 days before first simulation
  The Big Five Inventory-10 (BFI-10) measures the Big Five personality traits: Extraversion, Agreeableness, Conscientiousness, Emotional Stability, and Openness. Each question has five response options ranging in value from one to five (1= disagree strongly; 2= disagree a little; 3= neither agree or disagree; 4= agree a little; 5= agree strongly). To find the total raw score, sum the values of the response to each question for each of subscale (reverse code items 1,3,4,5 and 7). The lowest possible raw score is 10 and the highest possible raw score is 50. A score ranging from 2-10 is obtained by summing each factor individually. A higher score represents more of the concept being measured.
Rosenberg Self-Evaluation Scale (RSES) | 2 days before first simulation
  The Rosenberg Self-Evaluation Scale was used to measure the individual's global self-esteem and overall relationship to self. This questionnaire contains 10 items, five of which are worded positively and five negatively. Respondents rate their answers on a scale from 1 ('completely invalid') to 4 ('completely valid'). A total score, indicating the level of self-esteem, is obtained by summing all responses - a higher total score indicates a higher level of self-esteem.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Masaryk University, Brno, Bohunice, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dunton H, Leng O, Catlow J, Hancock J, Metcalf J. Stress and heart rate in high-fidelity training scenarios for undergraduate medical students. Future Hosp J. 2016 Jun 1;3(Suppl 2):s16. doi: 10.7861/futurehosp.3-2s-s16. No abstract available. PMID 31098245
- [Background] Peabody JE, Ryznar R, Ziesmann MT, Gillman L. A Systematic Review of Heart Rate Variability as a Measure of Stress in Medical Professionals. Cureus. 2023 Jan 29;15(1):e34345. doi: 10.7759/cureus.34345. eCollection 2023 Jan. PMID 36865953
- [Background] van Dulmen S, Tromp F, Grosfeld F, ten Cate O, Bensing J. The impact of assessing simulated bad news consultations on medical students' stress response and communication performance. Psychoneuroendocrinology. 2007 Sep-Nov;32(8-10):943-50. doi: 10.1016/j.psyneuen.2007.06.016. Epub 2007 Aug 6. PMID 17689196